CLINICAL TRIAL: NCT01864655
Title: A Phase Ib Multiple Ascending Dose Study of the Safety, Tolerability, and CNS Availability of AZD0530 in Alzheimer's Disease
Brief Title: Safety and Tolerability of AZD0530 (Saracatinib) in Alzheimer's Disease
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Stephen M. Strittmatter (Other)
Collaborators: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Sponsor-Investigator, Stephen M. Strittmatter, Professor of Neurology and Neurobiology, Yale University
Organization: Yale University (Other)
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1303011664; 1UH2TR000967-01 (NIH); 1R01NS084911-01 (NIH)
Record Dates: First submitted 2013-05-08; First posted 2013-05-29 (Estimated); Last update posted 2021-04-23 (Actual); Status verified 2021-04

CONDITIONS: Alzheimer's Disease
MeSH Terms: conditions — Alzheimer Disease | interventions — saracatinib

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Saracatinib group 1 (Experimental): This group will receive AZD0530 (saracatinib) experimental oral drug , once daily, for a duration of 4 weeks. Dosage is 50mg per day.
  Interventions: Drug: saracatinib
- Saracatinib group 2 (Experimental): Group 2 will receive saracatinib at a daily oral dose determined by the response to 50mg P.O. daily. Duration is 4 weeks.
  Interventions: Drug: saracatinib
- Saracatinib group 3 (Experimental): Group 3 will receive saracatinib at a dose determined by the response to 50mg P.O. daily, as well as dose given to group 2. Duration is 4 weeks.
  Interventions: Drug: saracatinib
- Placebo group 1-3 (Placebo Comparator): Subjects receiving saracatinib in groups 1-3 will be compared to subjects receiving daily, oral, placebo drug.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: saracatinib — oral drug given to experimental group
  Other Names: AZD0530
  Arms: Saracatinib group 1; Saracatinib group 2; Saracatinib group 3
Drug: Placebo — Placebo given to placebo group
  Arms: Placebo group 1-3

SUMMARY:
Alzheimer's disease is a devastating neurodegenerative disorder, for which there is currently no effective treatment to slow or halt progression. Beta amyloid peptide accumulates in the brains of those with Alzheimer's, and is thought to play a major role in triggering the dementia. The investigators recently characterized a molecular pathway by which ß-amyloid damages neurons, and showed that the protein termed Fyn kinase is crucial. Our data suggest that blocking Fyn will have a significant therapeutic benefit for Alzheimer's. Astra Zeneca has developed a blocker of Fyn and related kinases (AZD0530) for the treatment of cancer. Chronic AZD0530 administration is well tolerated in humans, and the investigators propose to test its potential as a novel Alzheimer's disease modifying therapy. This study will assess the safety and tolerability of AZD0530 in patients with Alzheimer's disease.

ELIGIBILITY:
Inclusion Criteria:

1. NIA-Alzheimer's Association core clinical criteria for probable AD 2. Age between 50-90 (inclusive). 3. MMSE score between 16 and 26 (inclusive) 4. Clinical Dementia Rating = 0.5, 1.0, or 2 5. Stability of permitted medications for 4 weeks. In particular, subjects may:

1. Take stable doses of antidepressants (if they are not currently depressed or do not have a history of major depression within the past 1 year).
2. Washout from psychoactive medication for at least 4 weeks prior to screening.
3. Cholinesterase inhibitors are allowable if stable for 12 weeks prior to screen. 6. Geriatric Depression Scale less than 6. 7. Study partner is available who has frequent contact with the subject (e.g. an average of 8 hours per week or more), and can accompany the subject to all clinic visits for the duration of the protocol.

   8. Visual and auditory acuity adequate for neuropsychological testing. 9. Good general health with no diseases expected to interfere with the study. 10. Subject is not pregnant, lactating, or of childbearing potential (i.e. women must be two years post-menopausal or surgically sterile).

   11. Modified Hachinski less than or equal to 4. 12. Completed six grades of education or has a good work history (sufficient to exclude mental retardation).

   13. Must speak English or Spanish fluently.

   Exclusion Criteria:
   1. Any significant neurologic disease other than AD, such as Parkinson's disease, multi-infarct dementia, Huntington's disease, normal pressure hydrocephalus, brain tumor, progressive supranuclear palsy, seizure disorder, subdural hematoma, multiple sclerosis, or history of significant head trauma followed by persistent neurologic defaults or known structural brain abnormalities
   2. Screening/baseline MRI scan with evidence of infection, infarction, or other focal lesions. Subjects with multiple lacunes or lacunes in a critical memory structure are excluded.
   3. Subjects that have any contraindications for MRI studies, including claustrophobia, the presence of metal (ferromagnetic) implants, or cardiac pacemaker will be excluded from the study.
   4. Major depression, bipolar disorder as described in DSM-IV within the past 1 year. Psychotic features, agitation or behavioral problems within 3 months, which could lead to difficulty complying with the protocol.
   5. History of schizophrenia (DSM IV criteria).
   6. History of alcohol or substance abuse or dependence within the past 2 years (DSM IV criteria).
   7. Any significant systemic illness or unstable medical condition, which could lead to difficulty complying with the protocol.
   8. Clinically significant abnormalities in B12 or TFTs that might interfere with the study.
   9. Residence in skilled nursing facility.
   10. Current use (within 30 days of screening) of specific psychoactive medications (e.g., typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity, etc.). Current use of warfarin.
   11. Investigational amyloid lowering therapies are prohibited two months prior to screening and for the duration of the trial. Other investigational agents are prohibited one month prior to screening and for the duration of the trial.
   12. Current or recent participation in any procedures involving radioactive agents, including current, past, or anticipated exposure to radiation in the workplace, such that the total radiation dose exposure to the subject in a given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1. This guideline is an effective dose of 5 rem received per year.

   7. Clinically significant or unstable medical condition, including uncontrolled hypertension, uncontrolled diabetes, or significant cardiac, pulmonary, renal, hepatic, endocrine, or other systemic disease in the opinion of the Investigator, may either put the patient at risk because of participation in the study, or influence the results, or the patient's ability to participate in the study.

   8. Clinically significant abnormalities in B12 or TFTs that might interfere with the study.

   9. Residence in skilled nursing facility. 10. Current use (within 30 days of screening) of specific psychoactive medications (e.g., typical neuroleptics, narcotic analgesics, antiparkinsonian medications, systemic corticosteroids, or medications with significant central anticholinergic activity, etc.). Current use of warfarin.

   11. Investigational amyloid lowering therapies are prohibited two months prior to screening and for the duration of the trial. Other investigational agents are prohibited one month prior to screening and for the duration of the trial.

   12. Current or recent participation in any procedures involving radioactive agents, including current, past, or anticipated exposure to radiation in the workplace, such that the total radiation dose exposure to the subject in a given year would exceed the limits of annual and total dose commitment set forth in the US Code of Federal Regulations (CFR) Title 21 Section 361.1. This guideline is an effective dose of 5 rem received per year.

   13. Current use (within 30 days of screening and throughout the protocol including the 2 week follow-up period) of the following medications: a) strong CYP3A4 inhibitors including: atazanavir, indinavir, ritonavir, saquinavir, nelfinavir, ketoconazole, itraconazole, clarithromycin, telithromycin, and nefazodone; b) strong CYP3A4 including: rifampicin, phenytoin, phenobarbital, and carbamazepine; c) certain CYP3A4 substrates including colchicine, cyclosporine, disopyramide, fluticasone, quinidine, vinblastine, vincristine. Patients taking sildenafil, tadalafil, and vardenafil will be advised to stop taking these medications for the duration of the trial.

   14. Neutropenia defined as absolute neutrophils count of <1,500/microliter. 15. Thrombocytopenia defined as platelet count <100x103/microliter. 16. Current blood clotting or bleeding disorder, or significantly abnormal PT or PTT at screening.

   17. Clinically significant abnormalities in screening laboratories, including Aspartate aminotransferase (AST) >1.5 times ULN; Alanine aminotransferase (ALT) > 1.5 times ULN; Total bilirubin >1.5 times ULN; Serum creatinine >2.0 times ULN.

   18. History of interstitial lung disease.

Ages: 50 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2013-07; Primary Completion 2014-03 (Actual); Study Completion 2014-11-06 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Adverse Events on AZD0530 | up to 4 weeks
  Patients will be followed closely for any adverse events. These include laboratory measurements, such as complete blood cell counts, basic metabolic panel, including renal function and electrolyte levels, coagulations factors, and liver function tests. These measures will be assessed weekly. Patients will have cognitive testing weekly, to ensure the absence of a prominent decline in function while on study drug. General daily function will be assessed, and any clinical symptoms, such as dizziness, headache or other symptoms will be addressed. All measures will be compared to baseline testing before drug therapy is started.
CNS availability of AZD0530 after oral dosing | 4 weeks
  Cerebrospinal fluid will be obtained at the end of the study to measure drug level. CSF will be obtained by a lumbar puncture.

SECONDARY OUTCOMES:
Effects of AZD0530 on cognitive function in patients with Alzheimer's disease | 4 weeks
  Study participants will undergo a standard cognitive battery, including the Alzheimer's Disease Assessment Scale - cognitive subscale (ADAS-cog), Alzheimer's Disease Cooperative Study - Activities of Daily living Inventory (ADCS-ADL), Clinical Dementia Rating - Sum of Boxes (CDR-SOB), Neuropsychiatric Inventory (NPI), and Mini-Mental State Examination (MMSE) at baseline, and at the conclusion of the study. Standard scores from the baseline test battery will be compared to the results at the end of the study to assess any change as a consequence of drug therapy.
Effect of AZD0530 on brain glucose metabolism in patients with Alzheimer's disease | 4 weeks
  A brain FDG-PET scan will be obtained at baseline, and again at the end of the study. Brain glucose metabolism will be assessed quantitatively, and the baseline pre-drug scan will be compared to the scan obtained after 4 weeks of drug/placebo therapy.

CONTACTS AND LOCATIONS:
Overall Officials: Haakon B Nygaard, MD, PhD, Principal Investigator — Yale University; Christopher van Dyck, MD, Principal Investigator — Yale University; Stephen M Strittmatter, MD, PhD, Principal Investigator — Yale University
Locations (1):
- Yale Alzheimer's Disease Research Unit, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Nygaard HB, Wagner AF, Bowen GS, Good SP, MacAvoy MG, Strittmatter KA, Kaufman AC, Rosenberg BJ, Sekine-Konno T, Varma P, Chen K, Koleske AJ, Reiman EM, Strittmatter SM, van Dyck CH. A phase Ib multiple ascending dose study of the safety, tolerability, and central nervous system availability of AZD0530 (saracatinib) in Alzheimer's disease. Alzheimers Res Ther. 2015 Apr 14;7(1):35. doi: 10.1186/s13195-015-0119-0. eCollection 2015. PMID 25874001